CLINICAL TRIAL: NCT01501916
Title: Effect of Vitamin D3 on Cardiovascular Risk Factors: a Randomized Trial in Human
Brief Title: Effect of Vitamin D3 on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Ulf Schlegelmilch, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0315668A
Record Dates: First submitted 2011-11-04; First posted 2011-12-30 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hypertensive Disease; Deficiency of Vitamin D3
MeSH Terms: conditions — Hypertension | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin d (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — daily dosage of 50 µg Vitamin D3 for 8 weeks
  Other Names: cholecalciferol
  Arms: vitamin d
Dietary Supplement: Placebo — daily intake of placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether a supplementation of Vitamin D3 can be used to reduce atherosclerotic risk factors.

DETAILED DESCRIPTION:
It is the objective of this study to investigate whether a supplementation with Vitamin D3 can be used to reduce atherosclerotic risk factors such as hypertension, inflammation and hyperlipidemia. The research question is whether Vitamin D3 can lower blood pressure in mildly hypertensive subjects who are naive to antihypertensive medication, whether Vitamin D reduces the level of systemic inflammation and whether Vitamin D3 has an effect on blood lipids.

major outcomes:

- decrease of systolic blood pressure in the treatment group in comparison with the placebo group

ELIGIBILITY:
Inclusion Criteria:

* human volunteers with mild hypertension

Exclusion Criteria:

* use of antihypertensive medication
* use of vitamin d or calcium supplements
* known renal, inflammatory or malignant diseases
* hypercalcemia or hypercalciuria
* participation in other clinical studies
* use of tanning booths during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
blood pressure | after 8 weeks of supplementation
  major outcome variable is the decrease oy systolic blood pressure in the treatment group in comparison with the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, Prof. Dr., Study Director — Institut für Agrar- und Ernährungswissenschaften